CLINICAL TRIAL: NCT01174368
Title: An Open-Label, Phase II Efficacy Trial of the Implantation of Mouse Renal Adenocarcinoma Cell-Containing Agarose-Agarose Macrobeads in the Treatment of Subjects With Castration-Resistant Prostate Cancer Resistant to Taxanes (Docetaxel, Cabazitaxel) and Evidence of Disease Progression on Androgen-axis Inhibition and/or Immunotherapy in the Form of Sipuleucel-T
Brief Title: Efficacy Trial of the Implantation of Mouse Renal Adenocarcinoma Macrobeads in Subjects With Castration-Resistant Prostate Cancer Resistant to Taxanes (Docetaxel, Cabazitaxel) and Evidence of Disease Progression on Androgen-axis Inhibition and/or Immunotherapy in the Form of Sipuleucel-T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1003010955
Record Dates: First submitted 2010-08-01; First posted 2010-08-03 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cancer macrobeads (Experimental): Cancer Macrobead placement in abdominal cavity
  Interventions: Biological: Cancer Macrobead placement in abdominal cavity

INTERVENTIONS:
Biological: Cancer Macrobead placement in abdominal cavity — 8 macrobeads per kilogram

SUMMARY:
This is a clinical research study of an investigational (FDA IND-BB 10091) treatment of subjects with castration-resistant prostate cancer resistant to Taxanes (docetaxel, cabazitaxel) and evidence of disease progression on androgen-axis inhibition and/or immunotherapy in the form of sipuleucel-T.

The treatment is being evaluated for its effect on tumor growth. It consists of the placement (implantation) of small beads that contain mouse renal adenocarcinoma cells (RENCA macrobeads). The cells in the macrobeads produce substances that have been shown to slow or stop the growth of tumors in experimental animals and veterinary patients. It has been tested in 31 human subjects with different types of cancers in a Phase I safety trial. Phase II studies in patients with colorectal, pancreatic or prostate cancers are in progress.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of prostate
* Evidence of metastasis
* Failed available therapies
* Resolution of any toxic effects of previous therapies
* Performance status (ECOG PS) 0-2
* Adequate hematologic, coagulation (INR 2-3max), hepatic and renal function
* Life expectancy of 12 months
* Agrees to contraceptive use while on study if sexually active
* Sign informed consent document

Exclusion Criteria:

* Any condition presenting an unacceptably high anesthetic or surgical risk
* HIV positive
* Cognitive impairment such as to preclude informed consent
* Other surgical treatment, chemotherapy and radiation within four weeks of baseline
* Inadequate hematologic, coagulation (INR >3), hepatic, renal function
* Hepatic blood flow abnormalities and/or large-volume ascites
* Concurrent cancer of any other type except skin cancer (excluding melanoma)
* History of allergic reactions to mouse antigens
* Active infection, congestive heart failure, unstable angina, serious cardiac arrhythmias, psychiatric illness, difficult social situations not permitting reliable participation, active bleeding

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry H Smith, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cancer Macrobeads
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: No analysis was performed due to small sample size. The one baseline participant withdrew voluntarily from the study after first implantation.
Arm/Group | Cancer Macrobeads
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Data was not collected.
Time Frame: 16 months
Population: Data was not collected.
Arm/Group | Cancer Macrobeads
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Metastases
Time Frame: 16 months
Population: Data was not collected. No statistical analysis was performed due to the sample size of one patient.
Arm/Group | Cancer Macrobeads
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Description: No data was collected.
Time Frame: 16 months
Population: Data was not collected.
Arm/Group | Cancer Macrobeads
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cancer Macrobeads
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cancer Macrobeads (N=1)
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Decreased appetite (General disorders) | 1
Diaphoresis (General disorders) | 1
Urinary urgency (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes